CLINICAL TRIAL: NCT01086592
Title: Effects of a Program of Physical Exercise and Electrotherapy on Muscle Strength in Subjects of the Fourth Age
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Pedro Rosado Calatayud/Physical Therapy Coordinator, CEU-Cardenal Herrera
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEU-UCH-87
Record Dates: First submitted 2010-03-09; First posted 2010-03-15 (Estimated); Last update posted 2010-07-05 (Estimated); Status verified 2010-06

CONDITIONS: Geriatric Assessment; Muscle Strength; Postural Balance; Body Mass Index
Keywords: Aged; Strength; Balance; Electrotherapy; Quality of life
MeSH Terms: interventions — Electric Stimulation Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Active Comparator)
  Interventions: Other: No intervention
- Strengthening exercise (Experimental): Strong progressive strengthening exercises of lower limbs.
  Interventions: Other: Strong progressive strengthening exercises of lower limbs
- Electrotherapy (Experimental): Neuromuscular Electrical Nerve Stimulation
  Interventions: Other: Electrotherapy
- Electrotherapy+weights (Experimental)
  Interventions: Other: Electrotherapy+weights

INTERVENTIONS:
Other: No intervention — Daily life activities
  Arms: Control
Other: Strong progressive strengthening exercises of lower limbs — Lower limb weight
  Arms: Strengthening exercise
Other: Electrotherapy — Neuromuscular Electrical Nerve Stimulation
  Arms: Electrotherapy
Other: Electrotherapy+weights — Superimposed Neuromuscular Electric Nerve Stimulation
  Arms: Electrotherapy+weights

SUMMARY:
The purpose of this study is to determine whether neuromuscular electrical stimulation, strengthening exercises, or combination of both over lower limbs are effective in the improvement of the stability fundamentally against falls, greater independence and, therefore, better quality of life in elderly over 75 years.

ELIGIBILITY:
Inclusion Criteria:

* Age above 75

Exclusion Criteria:

* Mental disorder
* Previous electrotherapy treatments
* Pacemakers
* Lower limbs prosthetics
* Major coronary diseases

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 118 (Actual)
Dates: Start 2010-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Functional Capacity | 3 months
  Berg's Scale, SF-36 test, 6 minute walking test, Barthel test, SPPB.

SECONDARY OUTCOMES:
Strength in lower limbs | 3 months
  Dinamometry, bioimpedancy.
Timed standing balance. Side by side, semi tandem, tandem stand and one-leg stand | 3 months
  Berg Scale, SPPB.
Maximum Gait Speed. Time to cover a 4 meter distance | 3 months
  Physical performance test
Body mass index | 3 months
  Bioimpedancy, ecography, lower limb perimeter.
Six-minute walking test | 3 months
  Physical performance test, assessing maximum distance covered during 6 minutes (assistance allowed if required).

CONTACTS AND LOCATIONS:
Overall Officials: Javier Romero, Dean, Study Director — Facultad Ciencias Salud CEU-UCH
Locations (1):
- CEU-Cardenal Herrera University, Moncada, Valencia, Spain

REFERENCES:
- [Background] Barry BK, Carson RG. The consequences of resistance training for movement control in older adults. J Gerontol A Biol Sci Med Sci. 2004 Jul;59(7):730-54. doi: 10.1093/gerona/59.7.m730. PMID 15304540
- [Background] Bax L, Staes F, Verhagen A. Does neuromuscular electrical stimulation strengthen the quadriceps femoris? A systematic review of randomised controlled trials. Sports Med. 2005;35(3):191-212. doi: 10.2165/00007256-200535030-00002. PMID 15730336
- [Background] Caggiano E, Emrey T, Shirley S, Craik RL. Effects of electrical stimulation or voluntary contraction for strengthening the quadriceps femoris muscles in an aged male population. J Orthop Sports Phys Ther. 1994 Jul;20(1):22-8. doi: 10.2519/jospt.1994.20.1.22. PMID 8081406
- [Background] Hunter GR, McCarthy JP, Bamman MM. Effects of resistance training on older adults. Sports Med. 2004;34(5):329-48. doi: 10.2165/00007256-200434050-00005. PMID 15107011
- [Background] Paillard T, Noe F, Passelergue P, Dupui P. Electrical stimulation superimposed onto voluntary muscular contraction. Sports Med. 2005;35(11):951-66. doi: 10.2165/00007256-200535110-00003. PMID 16271009
- [Derived] Benavent-Caballer V, Rosado-Calatayud P, Segura-Orti E, Amer-Cuenca JJ, Lison JF. Effects of three different low-intensity exercise interventions on physical performance, muscle CSA and activities of daily living: a randomized controlled trial. Exp Gerontol. 2014 Oct;58:159-65. doi: 10.1016/j.exger.2014.08.004. Epub 2014 Aug 15. PMID 25131453